CLINICAL TRIAL: NCT03130608
Title: Comparison of Inspiratory Muscle Training and Usual Care in Individuals Post-Liver Transplant
Brief Title: Inspiratory Muscle Training Post-Liver Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, David W. Mandel, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170229
Record Dates: First submitted 2017-03-16; First posted 2017-04-26 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Liver Disease Chronic; Muscle Weakness; Respiratory Insufficiency
Keywords: liver disease; transplant; muscle wasting; breathing exercise
MeSH Terms: conditions — Muscle Weakness; Respiratory Insufficiency; Liver Diseases; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): The experimental group will perform Inspiratory Muscle Training (IMT) using a THRESHOLD device, a simple hand held one way valve.
  In addition, the experimental group will gradually increase their activity as part of their usual care post-transplant.
  Interventions: Other: Inspiratory Muscle Training
- Usual Care (No Intervention): Receive the usual post-liver transplant care of gradually increase their activity.

INTERVENTIONS:
Other: Inspiratory Muscle Training — Subjects will breath through a hand held valve that has adjustable resistance to strengthen the muscles used for breathing. Subjects will perform the exercise approximately 20-30 minutes, twice a day for 8 weeks.
  Arms: Inspiratory Muscle Training

SUMMARY:
Individuals with chronic liver disease develop significant muscle wasting that remains post-liver transplant. The transplant surgery additionally challenges respiratory mechanics. Respiratory muscle strength has been measured to be impaired in individuals post liver transplant. This study proposes an 8 week intervention designed to increase respiratory muscle strength and pulmonary function that we hypothesize will correlate to improved functional performance and quality of life post-liver transplant.

Pre-test post-test design, that will randomize subjects into an experimental group that will receive the inspiratory muscle strengthening exercise in addition to usual post-liver transplant care and a control group that will only receive the usual post-transplant care.

Up to 50 subjects will be recruited from the Post-Liver Transplant Outpatient Clinic at the Miami Transplant Institute.

The subjects will have repeated measurements of respiratory muscle strength, pulmonary function, functional mobility performance, and quality of life at baseline, 4 weeks, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have undergone liver transplantation for chronic liver disease of any origin other than cancer.

Exclusion Criteria:

1. Severe cardiopulmonary disease such as recent Myocardial infarction, Congestive Heart Failure, Pulmonary edema, Chronic Obstructive Pulmonary Disease, and Asthma,
2. Severe osteoarthritis
3. Blindness
4. Wheelchair bound individuals
5. Individuals with neurological / neuromuscular disorders including but not limited to: cerebral vascular accident, Parkinsonism, Alzheimer's disease, dystonia, multiple sclerosis, and polio.
6. Severe Cognitive impairment where individuals cannot follow commands and are unable to sign informed consent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Maximal Inspiratory Pressure (MIP) at 4 weeks and 8 weeks. | Baseline, 4 weeks, and 8 weeks.
  MIP is a measure of inspiratory muscle strength . Inspiratory testing will be performed using a Micro Mouth Pressure Manometer. 92887) Measurements will be performed in the testing position with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
  Each measurement will be performed 3 times with the maximal score recorded.
Change from baseline Forced Expiratory Volume (FEV1) at 4 weeks and 8 weeks | Baseline, 4th week, and 8th week
  FEV1 is how much air can be exhaled during a forced exhalation at one second. Inspiratory testing will be performed using a Micro Mouth Pressure Manometer. 92887) Measurements will be performed in the testing position with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
  Each measurement will be performed 3 times with the maximal score recorded.
Change from baseline 6 Minute Walk Distance at 4 weeks and 8 weeks. | Baseline, 4 weeks, and 8 weeks
  In a 100ft. straight hallway the subject will walk back and forth, from one end to the other, as many times as they can in 6 minutes. The subject will have the option to rest at any time during the six minutes. The clock will keep running whether the subject is walking or resting. The subject will be provided standardized cues to prevent unequal encouragement. The distance walked over the 6 minutes will be recorded. Throughout the walking test, the investigator will be walking nearby to guard patient from loss of balance or fall.
Change from baseline 30 Second Chair Stand Repetitions at 4 weeks and 8 weeks. | Baseline, 4 weeks, and 8 weeks
  From a straight back chair the subject will come to a complete stand and then return to sitting with arms across chest. The number of times the subject can stand in 30 seconds will be recorded. The investigator will be standing nearby guarding the subject to protect from any loss of balance or fall.
Change from baseline Chronic Liver Disease Questionnaire (CLDQ) Score at 4 weeks and 8 weeks. | Baseline, 4 weeks, and 8 weeks
  This is a paper and pencil questionnaire consisting of 29 items in 6 domains: 1) Abdominal Symptoms 2) Activity: eating habits and movement of heavy objects 3) Emotional Function 4) Fatigue: perception of decreased energy and sleepiness 5) Systemic symptoms 6) Worry: concerns regarding disease progression and family. Summary scores for each domain range from 1(most impaired) to 7 (least impaired). All items refer to the previous 2 weeks. Higher scores indicate less impairment.
Change from baseline Karnovsky Performance Status Score at 4 weeks and 8 weeks. | Baseline, 4 weeks, and 8 weeks
  This is a paper pencil questionnaire measuring functional impairment. The questionnaire is divided into three groups for classifying patient's ability to work, to carry on normal activity, and to care for themselves. The groups are further divided into eleven categories covering all level so functioning from normal (100) to dead (0). The lower the Karnovsky score, the worse the functional ability and survival for most serious illness. The liver transplant team records this measure prior to transplant. We will obtained pre-transplant scores from medical record for use in correlational analysis. This measure will also performed at baseline and post-testing.
Change from baseline Sustained Maximal Inspiratory Pressure (SMIP) at 4 weeks and 8 weeks. | Baseline, 4 weeks, and 8 weeks
  SMIP will be measured from residual volume to total lung capacity representing single breath work/endurance. Inspiratory testing will be performed using a Micro Mouth Pressure Manometer. 92887) Measurements will be performed in the testing position with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
Change from baseline Inspiratory Duration (ID) at 4 weeks and 8 weeks | Baseline, 4 weeks, and 8 weeks
  ID is the inspiratory flow during maximal inspiration effort with an isokinetic like resistance from the mouthpiece. Inspiratory testing will be performed using a Micro Mouth Pressure Manometer. 92887) Measurements will be performed in the testing position with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
Change from baseline Maximal Expiratory Pressure (MEP) at 4 weeks and 8 weeks. | Baseline, 4 weeks, and 8 weeks
  MEP is a measure of expiratory muscle strength measured from total lung capacity. Inspiratory testing will be performed using a Micro Mouth Pressure Manometer. 92887) Measurements will be performed in the testing position with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
Change from baseline Forced Vital Capacity (FVC) at 4 weeks and 8 weeks. | Baseline, 4 weeks, 8 weeks.
  FVC is the total amount of air exhaled during a pulmonary function test. Expiratory testing will be performed using the Jones Satellite Spirometer (Jones Medical Instrument Company, Oakbrook, Illinois 65021) Measurements will be performed in the manner described using American Thoracic Society guidelines with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
  Each measurement will be performed 3 times with the maximal score recorded.
Change from baseline Forced Expiratory Flow (FEF25-75%) at 4weeks and 8 weeks. | Baseline, 4 weeks, 8 weeks.
  FEF25-75% is the flow rate at 25% to 75% of Forced Vital Capacity. Expiratory testing will be performed using the Jones Satellite Spirometer (Jones Medical Instrument Company, Oakbrook, Illinois 65021) Measurements will be performed in the manner described using American Thoracic Society guidelines with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
  Each measurement will be performed 3 times with the maximal score recorded.
Change from baseline Peak Expiratory Flow Rate (PEFR) at 4weeks and 8 weeks. | Baseline, 4 weeks, 8 weeks.
  PEFR is a measure of how fast a person can exhale. Expiratory testing will be performed using the Jones Satellite Spirometer (Jones Medical Instrument Company, Oakbrook, Illinois 65021) Measurements will be performed in the manner described using American Thoracic Society guidelines with subjects in the seated position and the trunk at a 90 degree angle to the hips. Subjects will wear a nose clip during testing.
  Each measurement will be performed 3 times with the maximal score recorded.

CONTACTS AND LOCATIONS:
Overall Officials: David W Mandel, PT, PhD, Principal Investigator — University of Miami Miller School of Medicine Department of Physical Therapy
Locations (1):
- Miami Transplant Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No